CLINICAL TRIAL: NCT06100341
Title: Developing Immersive Gamification Technology System for Rehabilitation Management of Pediatric Patients With Cerebral Palsy and Mobility Limitations (Phase 2 Trial)
Brief Title: ImGTS for Patients With Cerebral Palsy and With Mobility Limitations (Phase 2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augmented eXperience E-health Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AXEL0004
Record Dates: First submitted 2023-09-27; First posted 2023-10-25 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head-mounted display (HMD) (Experimental): The HMD system uses a commercially available virtual headset, the Oculus/Meta Quest 2, which allows a user to view a virtual environment in 360 degrees and to interact with the environment using hand-tracking technology (i.e., when a user's hand is projected into the virtual world to be used for interactions and gestures).
  Interventions: Other: Virtual reality
- Semi-cave automatic virtual environment (semi-CAVE) (Experimental): The semi-CAVE system uses projectors and projector screens to provide a 270-degree view of the virtual environment. These projectors are connected to a powerful workstation (desktop computer), which uses HTC Vive trackers and base stations to track user movements and interactions
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — A role-playing game set in a spaceship in outer space where a user will need to accomplish three activities to complete the game. These activities were designed based on typical therapy goals for children with cerebral palsy of improving balance, gross motor performance, walking speed, and functional mobility.

SUMMARY:
The proposed research project aims to answer the question "Are immersive technology systems effective in the rehabilitation management of pediatric patients with cerebral palsy and with mobility limitations?". The current study is the second of three phases, and it aims to create an immersive gamification technology system for the management of patients with cerebral palsy and with mobility disorders and to determine its clinical effectiveness, safety, and usability among children with mild to moderate cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-12 years old
* Able to walk without a mobility device with limited speed, balance, and/or coordination (equivalent to Gross Motor Function Classification System - Expanded and Revised (GMFCS) Level I or II)
* Can handle objects easily and successfully (equivalent to Manual Ability Classification System, MACS, Level I)
* Able to follow one-step instructions during BOTMP

Exclusion Criteria:

* Children with CP functioning at GMFCS Level III or higher
* Children who are totally dependent (i.e., those who require 100% assistance or support from another adult to complete tasks or for transfers or ambulation)
* Have had episodes of seizures or previously diagnosed as having epilepsy or are taking antiepileptic or seizure medications
* Have significant visual impairment
* Have hearing impairment requiring hearing aid
* Have a history of motion sickness
* Experience claustrophobia

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Balance will be assessed using Pediatric Balance Scale | Within one hour after completion of the sixth session
  The Pediatric Balance Scale is used to assess skills in functional balance among school-aged children. It rates a child's ability and records the time it takes for a child to maintain balance in different scenarios. Items are rated from 0 to 4, with a minimum score of 0 and a maximum score of 56. Changes are noted to be significant if the Pediatric Balance Scale score improvements are at least 0.79 points for the Pediatric Balance Scale-static scale, 0.96 points for the Pediatric Balance Scale-dynamic scale, and 1.59 points on the Pediatric Balance Scale-total scale.
Balance will be assessed using the Timed Up and Go in Children | Within one hour after completion of the sixth session
  Timed-Up and Go in Children is a timed test of functional dynamic balance where a child is tasked to stand up from a sitting position, walk 3 meters, turn and walk back, and sit down.
Gross motor performance will be assessed using the Bruininks-Oseretsky Test of Motor Proficiency (Second Edition; Short Form) | Within one hour after completion of the sixth session
  The Bruininks-Oseretsky Test of Motor Proficiency (Second Edition) is a comprehensive test of a child's fine and gross motor skills
Walking speed will be assessed using 10MWT | Within one hour after completion of the sixth session
  The 10-meter walk test (10MWT) assesses the walking speed of a child over a short distance
Functional ability will be assessed using Bruininks-Oseretsky Test of Motor Proficiency (Second Edition, Short Form) | Within one hour after completion of the sixth session
  The Bruininks-Oseretsky Test of Motor Proficiency (Second Edition, Short Form) is a comprehensive test of a child's fine and gross motor skills
Functional ability will be assessed using Timed-Up and Go in Children | Within one hour after completion of the sixth session
  Timed-Up and Go in Children is a timed test of functional dynamic balance where a child is tasked to stand up from a sitting position, walk 3 meters, turn and walk back, and sit down.
Incidence of virtual reality sickness symptoms will be assessed using the Virtual Reality Sickness Questionnaire | Immediately after each intervention, within an hour of completion of the virtual reality game
  The VRSQ will measure a participant's experience with the following symptoms: general discomfort, fatigue, eye strain, difficulty focusing, headache, fullness of head, blurring of vision, dizziness (when eyes are closed), and vertigo. Symptoms will be rated on a 4-point scale: 0 or None, 1 or Slight, 2 or Moderate, and 3 or Severe.
Usability of the virtual reality intervention will be assessed using the System Usability Scale | Immediately after each intervention, within an hour of completion of the virtual reality game
  The SUS is a 10-item questionnaire that is widely used in the evaluation of various kinds and aspects of technology. Each question has five response options ranging from 'Strongly agree' to 'Strongly disagree', which has a corresponding number value. Each response is added and multiplied by 2.5 to obtain the final score that ranges from 0 to 100. A SUS score above 68 is considered above average.
Usability of the virtual reality intervention will be assessed using a researcher usability checklist | Immediately after each intervention, within an hour of completion of the virtual reality game
  Usability will also be measured by the application's performance. Effectiveness will be measured in terms of task completion within a given time period, while efficiency will be measured in terms of ease of use of the controllers and the interface. Satisfaction will be determined through observation of participant reactions.

OTHER OUTCOMES:
Acceptability of the intervention will be qualitatively assessed based on the perceptions of patients, caregivers, and patient advocates | Within one week after completing virtual reality experience
  Acceptability will be measured among a small group of patients, caregivers, and patient advocates through an interview and a focus group discussion. More positive perceptions indicate a higher level of acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Eliza R. Aguila, PhD, Principal Investigator — University of the Philippines Manila
Locations (1):
- University of the Philippines College of Allied Medical Professions Immersive Technology Laboratory, Manila, National Capital Region, Philippines

REFERENCES:
- [Background] Aguila, M.E.R. et al. (2023). Application Design of a Virtual Reality Therapy Game for Patients with Cerebral Palsy. In: Krouska, A., Troussas, C., Caro, J. (eds) Novel & Intelligent Digital Systems: Proceedings of the 2nd International Conference (NiDS 2022). NiDS 2022. Lecture Notes in Networks and Systems, vol 556. Springer, Cham. https://doi.org/10.1007/978-3-031-17601-2_17
- [Background] Boque, J.C. et al. (2023). Moving in Space: Development Process Analysis on a Virtual Reality Therapy Application for Children with Cerebral Palsy. In: Kabassi, K., Mylonas, P., Caro, J. (eds) Novel & Intelligent Digital Systems: Proceedings of the 3rd International Conference (NiDS 2023). NiDS 2023. Lecture Notes in Networks and Systems, vol 784. Springer, Cham. https://doi.org/10.1007/978-3-031-44146-2_20